CLINICAL TRIAL: NCT03521193
Title: Migraine in Patients Undergoing PFO (Patent Foramen Ovale) Closure: Evaluation of a Platelet-associated Pathophysiologic Linking Mechanism
Brief Title: pLatelEts And MigRaine iN patEnt foRamen Ovale
Acronym: LEARNER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Daniela Trabattoni, MD, FACC, Centro Cardiologico Monzino
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCM769
Record Dates: First submitted 2018-04-16; First posted 2018-05-11 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-12

CONDITIONS: Platelet Aggregation, Spontaneous; Migraine With Aura; Patent Foramen Ovale
Keywords: Migraine;; PFO; platelet reactivity; aura
MeSH Terms: conditions — Platelet Aggregation, Spontaneous; Migraine with Aura; Foramen Ovale, Patent; Migraine Disorders; Epilepsy

STUDY DESIGN:
Intervention Model Description: Group 1: patients treated with PFO closure Group 2: Healthy subjects on Aspirin therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraine evaluation in PFO patients (Experimental): Patients symptomatic for migraine with/o aura and addressed to patent foramen ovale closure (Occlutech Figulla Flex II PFO occluder device) for a previous ischemic event, will receive dual antiplatelet therapy (DAPT) for 2 months after procedure and aspirin alone subsequently. Patients will undergo evaluation of platelet reactivity, serotonin and cytokines before PFO closure with a dedicated device and at 6 months follow-up and these results compared to those of a control, group of healthy subjects treated with aspirin alone
  Interventions: Device: patent foramen ovale closure
- healthy subjects on aspirin treatment (No Intervention): 12 healthy subjects on 100 mg aspirin daily will be compared to PFO patients in terms of platelet reactivity, serotonin and cytokines

INTERVENTIONS:
Device: patent foramen ovale closure — Pts undergoing PFO closure will receive 2-months of DAPT and 6 months of aspirin after patent foramen ovale (PFO) closure; they will be compared to healthy subjects on aspirin treatment
  Other Names: Occlutech Figulla Flex II PFO device; aspirin
  Arms: Migraine evaluation in PFO patients

SUMMARY:
Migraine is a common, chronic neurovascular disorder characterized by attacks of severe headache, autonomic nervous system dysfunction and, in some patients, aura, and disabling neurological symptoms. Worldwide, migraine prevalence is as high as 18% in the general population. Increased frequency of patent foramen ovale (PFO) in migraineurs was first reported in 1998 in a case-control study. Since then, others have described a 60% prevalence of PFO in patients suffering from migraine with aura. The presence of a right-to-left shunt (RLS) is thought to be a potent trigger of migraine attacks, although the mechanism is unknown. Moreover, PFO closure has correlated with improved migraine symptoms in several retrospective uncontrolled studies. The aim of this single-center, prospective study is to assess the impact of PFO closure on migraine attacks over time together with evaluation of potential predictive risk factors.

DETAILED DESCRIPTION:
The Study will evaluate the results of approximately 100 subjects from a single center study registered in this trial. Subjects who experienced transient ischemic attack (TIA) or stroke with a clinical indication to PFO closure and symptomatic for migraine with/o aura are considered for a migraine score analysis at baseline before PFO closure and during the subsequent follow-up (FU) at 6 and 12-months, together with lab evaluation for platelet reactivity tests (P selectin, Thromboxane B2), Prostaglandin E1 and 2 (PGE1, PGE2), serotonin, cytokines and prostaglandin PGE1 urinary metabolite run under aspirin therapy.

The research questions are as follows:

Does the presence of a large PFO have any impact on migraine with aura?

Do migraineurs with aura and PFO have higher biomarkers of platelet activation than control patients? and are they at higher risk of stroke and TIA recurrences based on high on clopidogrel platelet reactivity?

What is the effect of PFO severity on monthly migraine frequency and aura frequency?

What is the result of PFO closure in migraineur patients with PFO? Do Migraine with aura patients with large PFO have higher platelet activation and better migraine resolution after PFO closure?

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with more than 2 criteria:
* Previous Stroke or TIA (transient ischemic attack)
* positive MRI for ischemic events -
* PFO with a baseline R-L shunt > 10 microembolic signals (MES) and > 20 MES during/after Valsalva Manoeuver
* Atrial septal aneurysm (ASA) or residual Chiari network or Eustachian Valve
* positive Thrombophilic screening (MTHFR/prot C/Prot S)
* Ability to sign the informed consent for the study participation

Exclusion Criteria:

* Patients older than 70 years
* Paroxysmal Atrial fibrillation
* Carotid, vertebral or basilar artery stenosis> 50% on duplex imaging
* Inadequate temporal bone windows (signals) for transcranial Doppler insonation
* medication overuse headache
* history of cognitive dysfunction, epilepsy, brain injury
* use of continuous positive airway pressure (CPAP) within 6 months of study enrollment
* Left Ventricular Ejection Fraction (LVEF) < 30%
* Moderate/severe mitral valve regurgitation
* Known Allergy to aspirin
* Known allergy to nickel
* Severe chronic kidney disease (GFR < 30 ml/min)
* Beck depression inventory score > or= 29
* State-trait anxiety inventory score exceeding cut-off for are and sex

Keywords: PFO, migraine, migraine with aura, aura, platelets

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Trabattoni, MD, Principal Investigator — Centro Cardiologico Monzino, IRCCS
Locations (1):
- Centro Cardiologico Monzino, IRCCS, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trabattoni D, Brambilla M, Canzano P, Becchetti A, Teruzzi G, Porro B, Fiorelli S, Muratori M, Tedesco CC, Veglia F, Montorsi P, Bartorelli AL, Tremoli E, Camera M. Migraine in Patients Undergoing PFO Closure: Characterization of a Platelet-Associated Pathophysiological Mechanism: The LEARNER Study. JACC Basic Transl Sci. 2022 Apr 13;7(6):525-540. doi: 10.1016/j.jacbts.2022.02.002. eCollection 2022 Jun. PMID 35818509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at Centro Cardiologico Monzino, Milan, Italy between February 2018 and April 2020
Pre-assignment Details: After screening of 93 consecutive PFO patients suffering from migraine 15 were excluded due to unwillingness to sign the informed consent, absence of patent PFO at the invasive evaluation, intolerance to antiplatelet therapy. Finally, 78 pts were enrolled in the study and assigned to the PFO Arm; another arm included 12healthy subjects on Aspirin treatment
Groups:
- PFO and Migraine Pts: 93 consecutive patients addressed to PFO closure and suffering from migraine with aura were prospectively screened. 78 patients were enrolled in the study (T0)
- Healthy Subjects on Aspirin: 12 healthy subjects on ASA treatment were the control group for phase 2 study
Period: Overall Study
Arm/Group | PFO and Migraine Pts | Healthy Subjects on Aspirin
Started | 78 (enrolled on the PFO closure hospitalization) | 12
Completed | 62 (8 pts refused to continue the study; 8 patients were non compliant to ASA treatment) | 12
Not Completed | 16 | 0
Not completed — Withdrawal by Subject | 8 | 0
Not completed — non compliant to ASA treatment | 8 | 0

BASELINE CHARACTERISTICS:
Population: Final evaluation was performed on 62 patients. This group was compared to a control group (12 healthy subjects) on aspirin. Comparison was performed before PFO closure (T0) and during follow-up (T1) in terms of serotonin, platelet aggregation and activation markers and cell-associated procoagulant effect
Groups:
- PFO Patients Enrolled: We enrolled consecutive patients who met the inclusion criteria, symptomatic for migraine alone and Migraine with aura (MHA) patients.
  The leading indication to PFO closure was a previous TIA or stroke in 37 patients while an off-label indication was offered to 25 patients. These pts underwent PFO closure with the Occlutech Figulla device and treated with dual antiplatelet therapy (Aspirin 100 mg/day + Clopidogrel 75 mg/day), followed by aspirin 100 mg/day alone.
- Healthy Subjects: Healthy subjects on aspirin treatment by at least 15 days were the comparative group for platelet aggregation markers and activation markers, platelet procoagulant, circulating serotonin and cell-associated procoagulant potential
- Total: Total of all reporting groups
Arm/Group | PFO Patients Enrolled | Healthy Subjects | Total
Number analyzed (Participants) | 78 | 12 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12) | 41 (10) | 40.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 8 | 71
  Male | 15 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 78 | 12 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 78 | 12 | 90
Migraine [Number; unit: Migraine] — number of participants sffering from Migraine alone (MA)
  Migraine | 60 | 0 | 60
Migraine with aura (MHA) [Number; unit: Migraine with aura] — Number of patients suffering from Migraine with aura (MHA)
  Migraine with aura | 18 | 0 | 18
Patients finally evaluated [Number; unit: participants] — Population: 8 patients refused to continue the study ; 8 patients were not compliant to aspirin treatment, therefore final analysis was performed on 62 patients
  participants
    number analyzed (Participants) | 62 | 12 | 74
    (all) | 62 | 12 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change in Migraine Characteristics
Description: The evaluation in absolute numbers of patients fully responders, non-responders or with a moderate benefit on migraine symptoms after PFO Closure was performed
Time Frame: The outcome data were evaluated at 6-months and 12-months after PFO closure and compared to baseline
Population: Analysis performed only in PFO Group patients as not applicable to the control Healthy subjects group
Measure: Count of Participants; unit: Participants
Groups:
- Migraine Assessment After PFO Closure: Migraine symptoms evaluation after PFO closure
Arm/Group | Migraine Assessment After PFO Closure
Number analyzed (Participants) | 62
Participants
  Migraine : Complete Migraine Resolution | 43
  Migraine : Non-responders | 2
  Migraine Symptoms improvement | 17

2. Primary Outcome: Migraine Assessment by Anzola's Score
Description: The change in migraine severity, incidence and duration with or without aura as measured by the Anzola's score (The score is the expression of the sum of each corresponding value referring to migraine duration, frequency and the presence or absence of aura). The minimum value was 2 and the maximum 9; the higher the value, worse is the migraine classification.
  Anzola's score: Duration 0=No pain 1=<6 hours 2=6-12 hours 3=>12 hours Frequency 0=No pain 1=1-4/month 2=5-9/month 3=>10/month Aura 0=No aura
  1=Aura in ≥1 attack
Time Frame: Baseline, 6 months and 12-months after PFO closure
Population: Analysis performed only in PFO Group patients as not applicable to the control Healthy subjects group
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PFO Patients Enrolled: We enrolled consecutive patients who met the inclusion criteria, symptomatic for migraine alone and Migraine with aura (MHA) patients. Eight patients refused to continue the study and eight were non-compliant to antiplatelet therapy during the follow-up. .
  The leading indication to PFO closure was a previous TIA or stroke in 37 patients while an off-label indication was offered to 25 patients. These pts underwent PFO closure with the Occlutech Figulla device and treated with dual antiplatelet therapy (Aspirin 100 mg/day + Clopidogrel 75 mg/day), followed by aspirin 100 mg/day alone.
Arm/Group | PFO Patients Enrolled
Number analyzed (Participants) | 62
score on a scale
  Anzola's score @Baseline | 7.2 (1.68)
  Anzola's score@6-mos post PFO Closure | 1.09 (1.47)
  Anzola's score @12-mos post PFO closure | 1.1 (1.57)

3. Secondary Outcome: Platelet Activation (I)
Description: Platelet Thrombin generation potential in migraineurs and healthy subjects
Time Frame: baseline and 6 months after PFO closure
Measure: Mean (Standard Deviation); unit: min
Groups:
- PFO Patients: Evaluation of Platelet thrombin generation potential in PFO patients at T0
- Healthy Subjects: Evaluation of Platelet thrombin generation potential in HS
- PFO Patients at T1 (6 Mos): Evaluation of Platelet thrombin generation potential in PFO patients at T1 (6 mos)
Arm/Group | PFO Patients | Healthy Subjects | PFO Patients at T1 (6 Mos)
Number analyzed (Participants) | 62 | 15 | 62
min
  Lag Time | 26.9 (8.9) | 30.6 (7.2) | 32.2 (12.4)
  Time to peak | 32.1 (9.5) | 37.6 (10.2) | 37.8 (13)

4. Secondary Outcome: Platelet Activation (II)
Description: Platelet Thrombin generation Potential in Migraneurs and Healthy subjects
Time Frame: Baseline and 6 months after PFO closure
Population: Analysis of platelets' intrinsic characteristics including thrombin-formation capacity, the amount of thrombin and the kinetic rate (peak velocity)
Measure: Mean (Standard Deviation); unit: nMol/L/min
Groups:
- PFO Patients: Platelets kinetic rate (velocity index) at baseline, before PFO closure
- Healthy Subjects: Platelets kinetic rate (velocity index) in healthy subjects
- PFO Patients at T1 (6 Mos): Platelets kinetic rate (velocity index) at T1, six months after PFO closure
Arm/Group | PFO Patients | Healthy Subjects | PFO Patients at T1 (6 Mos)
Number analyzed (Participants) | 62 | 12 | 62
nMol/L/min | 29.1 (29) | 12.3 (10.9) | 17.9 (19.9)

5. Secondary Outcome: Platelet Activation (III)
Description: Platelets' endogenous thrombin generation potential in Migraneurs and Healthy subjects
Time Frame: baseline and six months after PFO closure
Measure: Mean (Standard Deviation); unit: nmol/L x min
Groups:
- PFO Patients at Baseline T0: Evaluation of Platelets' ETP (Endogenous Thrombin Potential) capacity before PFO closure
- Healthy Subjects: Evaluation of Platelets' ETP (Endogenous Thrombin Potential) capacity in HS on aspirin treatment
- PFO Patients at T1 (6 Mos): Evaluation of Platelets' ETP (Endogenous Thrombin Potential) capacity six months after PFO closure
Arm/Group | PFO Patients at Baseline T0 | Healthy Subjects | PFO Patients at T1 (6 Mos)
Number analyzed (Participants) | 62 | 12 | 62
nmol/L x min | 1038 (352) | 781 (319) | 797 (373)

6. Secondary Outcome: Platelet Activation (IV)
Description: Platelets' functional activity measured as the amount of thrombin generation
Time Frame: Baseline and six-months after PFO closure
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- PFO Patients at Baseline T0: Platelets' functional activity expressed as the amount of thrombin generated in PFO patients
- Healthy Subjects: Platelets' functional activity expressed as the amount of thrombin generated in HS on aspirin therapy
- PFO Patients at T1 (6 Mos): Platelets' functional activity expressed as the amount of thrombin generated six months after PFO closure
Arm/Group | PFO Patients at Baseline T0 | Healthy Subjects | PFO Patients at T1 (6 Mos)
Number analyzed (Participants) | 62 | 12 | 62
nmol/L | 115.2 (81.2) | 63.4 (41.8) | 77.2 (59.2)

7. Secondary Outcome: Platelet Aggregation (I)
Description: Platelet aggregation was measured on PAP-8 aggregometer (BioData). Briefly, PRP aliquots (250µL) were pipetted into a siliconized glass cuvette, stirred at 1200 rpm at 37°C and stimulated with arachidonic acid (1mM), collagen (2µg/ml), ADP (5µM), TRAP-6 (5µM). Light transmission was recorded for 5 min after stimuli addition and platelet aggregation was reported as maximal percentage of light transmission. Aspirin-treated patients were considered drug responders when platelet aggregation was less than 20% after arachidonic acid (1mM) stimulation.
Time Frame: baseline and 6 months after PFO Closure
Population: Patients were analysed at baseline before PFO closure, six months after procedure and compared to healthy subjects
Measure: Median (Inter-Quartile Range); unit: AUC (AU x min)
Groups:
- PFO Patients at T0: Median value of platelet aggregation in PFO patients at T0 (baseline)
- PFO Patients at T1: Median value of platelet aggregation in PFO patients at T1 (six months)
- Healthy Subjects: Median value of platelet aggregation in PFO patients in HS patients
Arm/Group | PFO Patients at T0 | PFO Patients at T1 | Healthy Subjects
Number analyzed (Participants) | 62 | 62 | 12
AUC (AU x min)
  ADP (5µM) | 153 [92.5 to 210] | 157 [92 to 216] | 187 [116 to 253]
  TRAP-6 (5µM) | 8.5 [5 to 14] | 8 [4 to 13] | 11 [9 to 27]
  Collagen (2µg/ml) | 62 [23.7 to 121.2] | 76.5 [30.2 to 139.5] | 104 [73 to 184]

8. Secondary Outcome: Clinical Outcomes
Description: Absence of TIA and stroke recurrences after PFO closure and during the follow-up
Time Frame: In hospital, six and 12 months follow-up
Population: Clinical evaluation of neurologic recurrences or death was performed during in-hospital stay and subsequent follow-up; Analysis performed only in PFO Group patients as not applicable to the control Healthy subjects group
Measure: Count of Participants; unit: Participants
Groups:
- PFO Patients Enrolled: We enrolled 62 consecutive PFO patients suffering from migraine, addressed to PFO closure. The leading indication to PFO closure was a previous TIA or stroke in 37 patients while an off-label indication was offered to 25 patients.
Arm/Group | PFO Patients Enrolled
Number analyzed (Participants) | 62
Participants
  In -hospital vascular complications | 1
  device malpositioning/embolization | 0
  Transient atrial fibrillation | 5
  TIA/stroke post PFO Closure | 0
  Recurrent TIAs /stroke @6 months FU | 0
  Recurrent TIAs /stroke @12 months FU | 0

ADVERSE EVENTS:
Time Frame: in -hospital, 6 months and 1 year
Description: Adverse event definitions were the same adopted by clinicaltrials.gov ; EVENTS WERE COLLECTED during clinical visit in-hospital and at follow-up
Groups:
- Migraine Evaluation in PFO Patients: Patients symptomatic for migraine with/o aura and addressed to patent foramen ovale closure (Occlutech Figulla Flex II PFO occluder device) for a previous ischemic event, will receive dual antiplatelet therapy (DAPT) for 2 months after procedure and aspirin alone subsequently. Clinical evaluation performed during in-hospital stay, at 6- and 12-months follow-up
- Healthy Subjects: control Healthy subjects group
Arm/Group | Migraine Evaluation in PFO Patients | Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/12
Other Adverse Events (participants affected / at risk) | 0/62 | 0/12

LIMITATIONS AND CAVEATS:
MHA may have a multifactorial etiology. The role of oxidative stress appears consistent and corroborated by the in vitro data. The effect of serotonin and oxidative stress was tested on platelets from healthy subjects and not from pts because the Sars-Cov-2 pandemic imposed restrictions on pts enrolment. Finally, the thrombin generation capacity of platelets and MVs were included after the study started to support the pro-coagulant phenotype evidenced by ad interim flow cytometry data analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT03521193/Prot_SAP_000.pdf